CLINICAL TRIAL: NCT01883180
Title: Dose Study of Antithymocyteglobulin in Haploidentical Hematopoietic Stem Cell Transplantation for Acute Graft-versus-host Disease Prophylaxis
Brief Title: ATG in Haploidentical HSCT for Acute Graft-versus-host Disease Prophylaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Southern Medical University, China (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Fujian Medical University Union Hospital (Other); Xiangya Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, the director of Department of Hematology, Nanfang Hospital and vice director of Institute of Hematology, Southern Medical University., Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-201304-K1
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Antithymocyte Globulin; Viral Infection
Keywords: haploidentical hematopoietic Stem Cell Transplantation; Antithymocyte globulin; viral infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATG 7.5mg/kg (Experimental): ATG 7.5mg/kg group refers to treatment with ATG in the total dose of 7.5mg/kg.
  Interventions: Drug: ATG
- ATG 10mg/kg (Experimental): ATG 10mg/kg group refers to treatment with ATG in the total dose of 10mg/kg.
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: ATG — ATG will be intravenously infused via a central venous catheter in 3 or 4 days, from day -4 or -3 until day -1. The other conditioning drugs administered before transplantation include cytosine arabinoside (Ara-C), busulfan (Bu),cyclophosphamide (Cy), Semustine(Me-CCNU), and ATG. All transplant recipients will receive cyclosporine A (CsA), mycophenolate mofetil(MMF), and short-term methotrexate for aGVHD prevention.

SUMMARY:
The purpose of this study is to compare the incidences of GVHD and viral infections in haploidentical hematopoietic stem cell transplant recipients receiving different dose of antithymocyte globulin (ATG) for acute graft-versus-host disease(aGVHD) prophylaxis. Our first objective was to investigate the optimal dose of ATG for aGVHD and second object was to evaluate the effect of different dose of ATG on post-transplant viral infection.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT)is the only therapeutic option for many hematological malignancies. Unfortunately, about 75% of patients who require allo-HSCT lack human leukocyte antigen (HLA)-matched donors. The alternative is hematopoietic stem cells from an HLA-mismatched family donor. However, this strategy, which is called haploidentical HSCT, may be associated with high risk of early death and severe GVHD.

Opportunistic infections are common complications after allo-HSCT. Due to the absence of effective preventive and therapeutic drugs for most viruses, viral infections has become one of the most important causes of death. The immunosuppression regimen including ATG has been shown effective to prevent severe GVHD in haploidentical HSCT. But this strategy delays immune reconstitution, and therefore increase the risk of viral infection.

The optimal dose of the different ATG preparations with respect to prevention of GvHD is not fully understood today. The total doses between 6 mg/kg to 15 mg/kg are effective for prevention of GVHD, but the dose above 10 mg/kg may increase the development of viral infection.

In this trial, we will focus on the incidence of aGVHD and viral infections in patients treated with 7.5mg/kg or 10mg/kg of ATG. The incidence of GVHD and viral infections will be compared between different dose arms.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 14-65 years
* Haploidentical hematopoietic stem cell transplant recipient
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2013-06; Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Epstein-Barr virus(EBV) viremia | 1 year
  Incidence of EBV viremia within 1 year

SECONDARY OUTCOMES:
Incidence of acute GVHD | 100 days
  Acute GVHD was graded according to standard criteria.
Incidence of EBV-associated diseases | 2 years
  the Incidence of EBV-associated end-organ diseases
Immune reconstitution | 1 year
  Immune reconstitution is performed every 3 months after transplantation.
Survival | 3 years
  Survival includes overall and disease-free survival within 2 years after transplantation.
Incidence of chronic GVHD | 2 years
  Chronic GVHD was assessed in patients alive after day 100.
Incidence of cytomegalovirus(CMV) viremia | 1 year
  Incidence of CMV viremia within 1 year
Incidence of CMV-associated diseases | 2 years
  the Incidence of CMV-associated end-organ diseases

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ottinger HD, Ferencik S, Beelen DW, Lindemann M, Peceny R, Elmaagacli AH, Husing J, Grosse-Wilde H. Hematopoietic stem cell transplantation: contrasting the outcome of transplantations from HLA-identical siblings, partially HLA-mismatched related donors, and HLA-matched unrelated donors. Blood. 2003 Aug 1;102(3):1131-7. doi: 10.1182/blood-2002-09-2866. Epub 2003 Apr 10. PMID 12689945
- [Background] Bacigalupo A, Lamparelli T, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Barbanti M, Sacchi N, Van Lint MT, Bosi A. Antithymocyte globulin for graft-versus-host disease prophylaxis in transplants from unrelated donors: 2 randomized studies from Gruppo Italiano Trapianti Midollo Osseo (GITMO). Blood. 2001 Nov 15;98(10):2942-7. doi: 10.1182/blood.v98.10.2942. PMID 11698275
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189
- [Derived] Fan M, Wang Y, Lin R, Lin T, Huang F, Fan Z, Xu Y, Yang T, Xu N, Shi P, Nie D, Lin D, Jiang Z, Wang S, Sun J, Huang X, Liu Q, Xuan L. Haploidentical transplantation has a superior graft-versus-leukemia effect than HLA-matched sibling transplantation for Ph- high-risk B-cell acute lymphoblastic leukemia. Chin Med J (Engl). 2022 Apr 20;135(8):930-939. doi: 10.1097/CM9.0000000000001852. PMID 35467818
- [Derived] Yu S, Huang F, Fan Z, Xuan L, Nie D, Xu Y, Yang T, Wang S, Jiang Z, Xu N, Lin R, Ye J, Lin D, Sun J, Huang X, Wang Y, Liu Q. Haploidentical versus HLA-matched sibling transplantation for refractory acute leukemia undergoing sequential intensified conditioning followed by DLI: an analysis from two prospective data. J Hematol Oncol. 2020 Mar 12;13(1):18. doi: 10.1186/s13045-020-00859-5. PMID 32164760
- [Derived] Lin R, Wang Y, Huang F, Fan Z, Zhang S, Yang T, Xu Y, Xu N, Xuan L, Ye J, Sun J, Huang X, Liu Q. Two dose levels of rabbit antithymocyte globulin as graft-versus-host disease prophylaxis in haploidentical stem cell transplantation: a multicenter randomized study. BMC Med. 2019 Aug 12;17(1):156. doi: 10.1186/s12916-019-1393-7. PMID 31401973